CLINICAL TRIAL: NCT02128204
Title: The Safety and Efficacy of Using HYADERMIS LA for Wrinkle Correction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SciVision Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RDCT-YDL
Record Dates: First submitted 2014-04-02; First posted 2014-05-01 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Pain; Nosalabial Folds Correction
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HYADERMIS LA Facial Dermal Implant (Experimental): Subjects will be randomly assigned to receive experiment treatment, lidocaine contained hyaluronate facial dermal filler, in one side of the face.
  Interventions: Device: lidocaine contained hyaluronate facial dermal filler
- Hya-Dermis Facial Dermal Implant (Active Comparator): Subjects will be randomly assigned to receive control treatment, hyaluronate facial dermal filler, in one side of the face.
  Interventions: Device: hyaluronate facial dermal filler

INTERVENTIONS:
Device: lidocaine contained hyaluronate facial dermal filler — HYADERMIS LA Facial Dermal Implant contains 20 mg/ml hyaluronate and 0.3 % lidocaine.
  Other Names: HYADERMIS LA Facial Dermal Implant
  Arms: HYADERMIS LA Facial Dermal Implant
Device: hyaluronate facial dermal filler — Hya-Dermis Facial Dermal Implant contains 20 mg/ml hyaluronate.
  Other Names: Hya-Dermis Facial Dermal Implant
  Arms: Hya-Dermis Facial Dermal Implant

SUMMARY:
The study is a double-blind, randomized, within-subject controlled, 2-armed, single-centre study sponsored by SciVision Biotech Inc. and approved by Yuan's General Hospital Institutional Review Board. The aim of this post-marketing study is to evaluate the safety and efficacy of HYADERMIS LA facial dermal implant for the improvement of nasolabial folds.

The study was estimated to be held half to one year including a 0-2 weeks screening period, a day of treatment, and follow-up at week 1 and 2. Patient informed consent forms will be obtained before volunteers enter screening period. If the volunteers meet all the criteria, they will be given a number to replace their name in the study. The participants will be randomised assigned to receive experiment treatment, HYADERMIS LA, in one side of nasolabial folds and control treatment, Hya-Dermis, in the other side of the face. The safety assessment evaluated any recorded adverse events following the device treatments either by blinded evaluator or subjects. The effectiveness of the treatment devices will be assessed by using photographic assessment, nasoalabial folds severity scale, global aesthetic improvement scale, and pain visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* Be 25 to 60 years of age and of any sex who is willing to receive nasolabial folds correction by intradermal injection procedures
* Have approximately symmetrical nasolabial folds with a nasolabial folds severity grade of 2-4 and the grade difference between two sides is less than 1
* Agree to refrain from undergoing invasive aesthetic treatments in the injective areas 12 months after the injections
* Agree to refrain from undergoing other physical or chemical aesthetic treatments in the injective areas 3 months after the injections
* If female of child-bearing potential, not be breastfeeding, have a negative urine pregnancy test on the treatment day and agree to use any approved contraceptives or medically acceptable method of birth control throughout the study
* Have ability to understand and comply with the study requirements, and provide the written informed consent prior to any procedures

Exclusion Criteria:

* Have history or active dermal diseases, inflammation, or any related disease
* Had permanent or semi-permanent implantation on nasolabial areas
* Had invasive aesthetic treatments or surgeries history 6 months before the treatments
* Had physical or chemical aesthetic treatments 1 months before the study starts
* Have history of coagulation defect diseases and still take aspirin, anticlotting, or blood activating medications 1 week before the treatments
* Have Adams-Stokes syndromes, wolff-prkinson-white syndromes, severe sinus node, the atrioventricular node dysfunction, or the blocked ventricular
* Have a known history of allergic reactions like hypersensitivity to hyaluronic acid
* Have a known history of allergic reactions like hypersensitivity to lidocaine or other anaesthetics
* Have poor compliance with the study or follow-up schedule

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Adverse events report | From the date of treatment to 14 days
  Any adverse events and abnormal physical parameters or reports occurred and disappeared should be monitored throughout the trial. The records should be assessed and keep on track of the severity of individual adverse events and correlation with the treatment. Severity assessment: To assess the level of severity by rating 0 (none), 1 (mild), 2 (median), and 3 (sever). Correlation assessment: Physicians evaluate the impact of adverse events for each individual and determine their causality of the treatment, giving score 0 (no correlated), 1 (low correlated), 2 (suspected correlated), 3 (most likely correlated ). Subjects will be given a medical diary after the treatment to record any adverse event and report to a physicians. Physicians keep following up adverse events until the symptoms stabilised.
Pain Visual Analog Scale | participants will be followed for the duration of treatment, an expected average of 10 minutes
  A quantification of the severity of pain experienced by the participants during the treatment. A scale of 100 mm horizontal line will be labeled by subjects to assess pain on both sides of the injected areas during the treatment. The one on the scale's extreme left (0) represents painless while the one on the extreme right (100) is set as the most pain could be imagined by subjects.

SECONDARY OUTCOMES:
Nasolabial folds severity scale | From the baseline, 30 minutes post-treatment, and every follow-up at 1 and 2 weeks
  Based on Skin Aging Altas: Volume 2, Asian type photographs, taking gender and nasolabial folds into consideration to quantify the degree of nosalabial folds severity. A validated 8-point photographic scale scored the severity grade from 0 (absent) 7 (extreme) will be used to assess the severity.
Global aesthetic improvement scale | 30 minutes post-treatments and follow-ups at 1 and 2 weeks
  To quantify the level of overall aesthetic improvement and so giving a scale from 1 (worse), 2 (no change), 3 (improved), and 4 (much improved), and 5 (very much improved).
Pain Visual Analog Scale | 15, 30, 45, and 60 minutes post-treatment
  A quantification of the severity of pain experienced by the participants after the treatment. A scale of 100 mm horizontal line will be labeled by subjects to assess pain on both sides of the injected areas at 15, 30, 45, and 60 minutes post-treatment. The one on the scale's extreme left (0) represents painless while the one on the extreme right (100) is set as the most pain could be imagined by subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Hong Liu, M.D., Principal Investigator — Department of Dermatology, Yuan's General Hospital
Locations (1):
- Aesthetic Center of Yuan's General Hospital, Kaohsiung City, Taiwan